CLINICAL TRIAL: NCT00144079
Title: Phase 3 Trial of Adjuvant External Beam Radiotherapy for Locally Invasive Differentiated Thyroid Carcinoma
Brief Title: Multicenter Study Differentiated Thyroid Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSDS; Deutsche Krebshilfe 70-2294
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2006-05-09 (Estimated); Status verified 2005-09

CONDITIONS: Thyroid Neoplasms
Keywords: Differentiated thyroid carcinoma; radiotherapy; radioiodine therapy; thyroidectomy
MeSH Terms: conditions — Thyroid Neoplasms

INTERVENTIONS:
Procedure: external beam radiotherapy

SUMMARY:
The trial examines the clinical benefit of adjuvant external beam radiotherapy (RTx) for locally invasive differentiated carcinoma (TNM stages pT4 pN0/1/x M0/x; 5th ed. 1997) of the thyroid gland (DTC). Patients are treated with surgery (thyroidectomy and lymphadenectomy), radioiodine therapy (RIT) to ablate the thyroid remnant tissue, and TSH-suppressive L-thyroxine therapy with or without RTx after documented elimination of cervical I-131 uptake.

DETAILED DESCRIPTION:
MSDS was designed as a comprehensive cohort trial with randomization and observation arms. Patients are enrolled at the time of the first ablative radioiodine therapy (RIT). Inclusion criteria are papillary or follicular DTC pT4 pN0/1/x M0/x, age between 18 (incl.) and 70 years (excl.) at the time of initial surgery, completion of primary surgical therapy with R0 (no tumor residues) or R1 (microscopic residues) resection, Karnofsky index of at least 70 %, freedom from distant metastases at the time of initial radioiodine therapy (RIT), and informed patient consent. Criteria for exclusion are secondary malignancy except basalioma, pregnancy, serious general disease, serious psychiatric disorder, inability to give informed consent, previous RTx and recurrence of previous DTC. From 2003, the first inclusion criterion was changed into DTC pT3/4 pN0/1/x M0/x to reflect the 2002 revision of the TNM staging system.

The treatment protocol is in accordance with current guidelines in Germany and includes total thyroidectomy (TT) with central lymphadenectomy (LNA), RIT to ablate the thyroid remnant, and TSH-suppressive therapy with L-thyroxine (TSH < 0.1 mU/l). RIT is administered under endogenous TSH-stimulation after 4 weeks' cessation of L-thyroxine using standard activities of 1-4, and 1-2, GBq I-131 in patients with a 24-h-I-131 uptake below 10 % and 10-20 %, resp., or individual dosimetry aiming for at least 300 Gy in the thyroid remnant. If scintigraphic I-131 uptake by the thyroid remnant persists at whole-body scintigraphy (at least 200 MBq; at least 48 h) 3 months after RIT, a second fraction of RIT is given with 4-10 GBq.

Patients who consented to randomization at centers actively taking part in randomization were randomized to treatment arms A (additional adjuvant RTx) and B (no RTx) 3 months after initial RIT after confirmation of the histological diagnosis by the reference pathologist and when distant metastases had been excluded by means of serum thyroglobulin (Tg), WBS (s. a.) and a native thoracic computed tomogram (CCT). Randomization was stratified according to histological type (papillary v. follicular), nodal status (pN0/1/x), and participating center, and performed by an operator-independent randomization routine embedded in the database. The remaining patients were assigned to arms A and B by the participating centers.

RTx is begun after documented elimination of cervical I-131 uptake in a I-131 WBS 3 months after the last fraction of ablative RIT. RT includes the thyroid bed (in unilateral tumors only the affected side) with a dose of 59.4 Gy and 66.6 Gy after R0 and R1 resection, resp., and the regional lymph nodes of the neck and upper mediastinum including the posterior cervical chain from the mandible and mastoid process to the tracheal bifurcation with a dose of 50.4 Gy and 54.0 Gy in pN0 and pN1/x disease, resp. Fractionation is conventional (1.8 Gy/d 5 days a week). 3-D planning according to IRCU 50 is mandatory.

Patient follow-up includes, as a minimum, out-patient appointments with cervical ultrasound and measurement of serum TSH, hTG, anti-Tg antibodies and a blood count 2 and 8 months after each RIT or WBS, and a WBS (with at least 200 MBq over at least 48 h) under endogenous TSH-stimulation 3 and 12 months after ablative RIT and then at 24-month intervals. FDG-PET and other imaging modalities can be performed if needed. At each follow-up appointment, RTx toxicity is recorded according to RTOG criteria and quality of life by the QLQ-C30 questionnaire (v. 3.0 German) of the EORTC.

ELIGIBILITY:
Inclusion Criteria:

* papillary or follicular thyroid carcinoma pT4 pN0/1/x M0/x
* completion of primary surgical therapy with R0 (no tumor residues) or R1 (microscopic residues) resection
* Karnofsky index > 70 %
* freedom from distant metastases at the time of initial radioiodine therapy
* informed patient consent

Exclusion Criteria:

* secondary malignancy except basalioma
* pregnancy
* serious general disease
* serious psychiatric disorder
* inability to give informed consent
* previous RTx
* recurrence of previous thyroid cancer

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2000-01; Study Completion 2010-01

PRIMARY OUTCOMES:
time to local or distant failure
cancer-related mortality

SECONDARY OUTCOMES:
acute toxicity of radiotherapy (RTOG)
chronic toxicity of radiotherapy (RTOG)
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Otmar Schober, Prof MD PhD, Study Chair — Department of Nuclear Medicine, Münster University Hospital, Münster, Germany; Henning Dralle, Prof MD, Study Director — Dept. of General Surgery, University Halle-Wittenberg, Halle, Germany; Normann Willich, Prof MD, Study Director — Department of Radiooncology, Münster University Hospital, Münster, Germany; Martin Biermann, MD, Study Director — Dept. of Nuclear Medicine, Münster University Hospital; Burkhard Riemann, MD PhD, Study Director — Dept. of Nuclear Medicine, Münster University Hospital; Andreas Schuck, MD PhD, Study Director — Dept. of Radiooncology, Münster University Hospital
Locations (10):
- Austria (2):
  - Department of Nuclear Medicine, Linz
  - Department of Nuclear Medicine, Wien University Hospital, Vienna
- Germany (7):
  - Department of Nuclear Medicine, Cologne University, Cologne
  - Department of Nuclear Medicine, University Halle-Wittenberg, Halle
  - Department of Nuclear medicine, Saarland University, Homburg/Saar
  - Department of Nuclear Medicine, Münster University Hospital, Münster
  - Department of Nuclear Medicine, Katharinen-Hospital, Stuttgart
  - Department of Nuclear Medicine, Helios-Klinikum Wuppertal, Wuppertal
  - Department of Nuclear Medicine, Würzburg University, Würzburg
- Department of Nuclear Medicine, Zürich University Hospital, Zurich, Switzerland

REFERENCES:
- [Background] Puskas C, Schober O. [Adjuvant percutaneous radiation of locally advanced papillary and follicular thyroid carcinoma: reflections for the necessity of a prospective multicenter study]. Nuklearmedizin. 1999;38(8):328-32. German. PMID 10615667
- [Background] Biermann M, Schober O; Multizentrische Studie Differenziertes Schilddrusenkarzinom Studiengruppe. [How many high-risk patients with differentiated thyroid cancer need a "Tumor Center" per year?]. Nuklearmedizin. 2002 Apr;41(2):61-2. No abstract available. German. PMID 11989299
- [Background] Biermann M, Schober O. GCP-compliant management of the Multicentric Study Differentiated Thyroid Carcinoma (MSDS) with a relational database under Oracle 8i. Inform Biom Epidemiol Med Biol 33:441-59, 2002
- [Background] Biermann M, Pixberg M, Schuck A, Willich N, Heinecke A, Schober O. External beam radiotherapy. An evidence-based review. In: Biersack H-J, Grünwald F, eds. Thyroid cancer. Heidelberg: Springer; 139-61, 2005.
- [Result] Biermann M, Pixberg MK, Schuck A, Heinecke A, Kopcke W, Schmid KW, Dralle H, Willich N, Schober O. Multicenter study differentiated thyroid carcinoma (MSDS). Diminished acceptance of adjuvant external beam radiotherapy. Nuklearmedizin. 2003 Dec;42(6):244-50. PMID 14668957
- [Result] Schuck A, Biermann M, Pixberg MK, Muller SB, Heinecke A, Schober O, Willich N. Acute toxicity of adjuvant radiotherapy in locally advanced differentiated thyroid carcinoma. First results of the multicenter study differentiated thyroid carcinoma (MSDS). Strahlenther Onkol. 2003 Dec;179(12):832-9. doi: 10.1007/s00066-003-1158-1. PMID 14652672
- [Result] Biermann M, Pixberg MK, Dorr U, Dietlein M, Schlemmer H, Grimm J, Zajic T, Nestle U, Ladner S, Sepehr-Rezai S, Rosenbaum S, Puskas C, Fostitsch P, Heinecke A, Schuck A, Willich N, Schmid KW, Dralle H, Schober O; MSDS study group. Guidelines on radioiodine therapy for differentiated thyroid carcinoma: impact on clinical practice. Nuklearmedizin. 2005;44(6):229-34, 236-7. PMID 16400382
- [Derived] Vrachimis A, Wenning C, Gerss J, Dralle H, Vaez Tabassi M, Schober O, Riemann B; MSDS study group. Not all DTC patients with N positive disease deserve the attribution "high risk". Contribution of the MSDS trial. J Surg Oncol. 2015 Jul;112(1):9-14. doi: 10.1002/jso.23948. Epub 2015 Jun 12. PMID 26074402
- [Derived] Riemann B, Kramer JA, Schmid KW, Dralle H, Dietlein M, Schicha H, Sauerland C, Frankewitsch T, Schober O; MSDS study group. Risk stratification of patients with locally aggressive differentiated thyroid cancer. Results of the MSDS trial. Nuklearmedizin. 2010;49(3):79-84. doi: 10.3413/nukmed-0302. PMID 20505894
- [Derived] Biermann M, Pixberg M, Riemann B, Schuck A, Heinecke A, Schmid KW, Willich N, Dralle H, Schober O; MSDS study group. Clinical outcomes of adjuvant external-beam radiotherapy for differentiated thyroid cancer - results after 874 patient-years of follow-up in the MSDS-trial. Nuklearmedizin. 2009;48(3):89-98; quiz N15. doi: 10.3413/nukmed-0221. Epub 2009 Mar 23. PMID 19322503